CLINICAL TRIAL: NCT01298245
Title: Genetic Association Studies of Diabetic Retinopathy (1): Vanguard Phase
Brief Title: Genetic Association of Diabetic Retinopathy-1
Acronym: DMR-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Yen Tjing Ling Medical Foundation (Unknown)
Responsible Party: Principal Investigator, vghtpe user, Attending physician, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 201008023GB; CI-99-1 (Other Grant/Funding Number: Yen Tjing Ling Medical Foundation)
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Diabetes; Diabetic Retinopathy
Keywords: diabetes; diabetic retinopathy; Chinese; gene; associations
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The participants will receive fasting blood sampling for the measurements of glucose, HbA1c, lipid profile, and biochemistry. An additional 10 ml blood sample will be taken for DNA extraction from buffy coat. Early morning urine samples will also be collected for evaluation of overt proteinuria by a dipstick method.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: diabetic retinopathy: Patients with diabetes who have received ophthalmic fundus examination within 6 months before the study and those with known positive results of diabetic retinopathy
- Control: no diabetic retinopathy: Patients with diabetes who have received ophthalmic fundus examination within 6 months before the study and those without known positive results of diabetic retinopathy

SUMMARY:
The primary purpose of the study is to investigate allele frequencies of candidate genes in Chinese diabetic patients with or without known diabetic retinopathy. Two hundred Chinese diabetic patients, aged between 20 - 75 years old, who have received ophthalmic fundus examination (either by an ophthalmoscope or fundus camera) within 6 months before the study will be recruited for the study. Each subject will receive anthropometric and blood pressure measurements. Then, fasting blood samples will be taken for the measurements of glucose, HbA1c, lipid profile, and biochemistry. An additional 10 ml blood sample will be taken for DNA extraction from buffy coat. Meanwhile, the participant will receive structural questionnaires for demography, personal history, medical history and concomitant medication. Single nucleotide polymorphisms (SNPs) in candidate genes and in targeted chromosome regions will be genotyped by using the ABI TaqMan assays. The differences in the distribution of genotypes and alleles between the study groups will be analyzed using appropriate statistical methods. Through the study, the investigators hope to build up a platform for future large-scale genetic studies of diabetic retinopathy. The investigators also hope to set up priority of candidate loci for future studies.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is one of the most frequent microvascular complications of diabetes (DM). Current guidelines recommend that patients with DM should receive ophthalmic fundus examination annually. DR poses a serious threat to the health of millions patients who have DM. Nowadays, DR has become the leading cause of new cases of visual impairment and blindness among adults.

Genetic factors are likely to account for the susceptibility to DR for the differences in DR incidence between individuals with diabetes. Familial aggregation studies showed that increased risk of severe DR was noted among family members with diabetes with moderate heritability of DR risk. Racial and ethnic differences in the prevalence of DR may also explain some parts of influence of genetic or environmental/cultural risk factors. There were over 30 candidate genes involved in metabolic mechanisms and functional pathways associated with DR. However, consistent associations between candidate genes and DR have yet been identified. The current study is designed to build up a working platform for future large-scale genetic studies of diabetic retinopathy. The investigators also hope to set up priority of candidate loci for future researches.

In the present study, the investigators plan to recruit 200 Chinese patients with DM who have received ophthalmic fundus examination (either by an ophthalmoscope or fundus camera) within 6 months before the study. Each subject will receive anthropometric and blood pressure measurements. Then, fasting blood samples will be taken for the measurements of glucose, HbA1c, lipid profile, and biochemistry. An additional 10 ml blood sample will be taken for DNA extraction from buffy coat. Single nucleotide polymorphisms (SNPs) in candidate genes and in targeted chromosome regions will be genotyped by using the ABI TaqMan assays. The differences in the distribution of genotypes and alleles between the study groups will be analyzed using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DM, diagnosed by the 2010 American Diabetes Association diagnosis criteria.
* Men or women.
* Aged 20 ~ 75 years old (inclusive).
* Who have received ophthalmic fundus examination within 6 months before the study: either (1)by an ophthalmoscope or fundus camera (results reviewed by a qualified physician), or (2)the ophthalmoscopic examination being performed by an ophthalmologist.
* Willing to participate in the study by signing an informed consent.

Exclusion Criteria:

* Women in pregnancy.
* No document to verify the results of the ophthalmic fundus examination requiring for the inclusion.
* History of mental incapacity or language barriers that may preclude adequate understanding or cooperation in the study.
* Current or concomitant illness that would interfere with the subject's ability to perform the study or that would confound the study results, judged by the investigation physicians.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with DM who have received ophthalmic fundus examination within 6 months before the study, either with or without diabetic retinopathy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The differences in the distribution of candidate genotypes and alleles between the study groups | 12 months
  Patients with diabetes who have received ophthalmic fundus examination within 6 months before the study. The eligible participants will be grouped by the results of prior fundus examination: those with known history of diabetic retinopathy; those without known history of diabetic retinopathy.

SECONDARY OUTCOMES:
the frequencies of haplotypes of different single nucleotide polymorphisms | 12 months
  We will estimate the frequencies of haplotypes of different single nucleotide polymorphisms, calculate linkage disequilibrium between single nucleotide polymorphisms, and conduct haplotype analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Chii-Min Hwu, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan